CLINICAL TRIAL: NCT00923988
Title: Acute Effects of Short-term Exposure to Secondhand Smoke on Platelet Activation and Endothelial Function
Brief Title: Effect of Passive Smoking on Platelet Function and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Graubünden (Other)
Responsible Party: Walter H. Reinhart, Head of the Department of Internal Medicine, Kantonsspital Graubuenden, Kantonsspital Graubuenden, Chur, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHS-EF
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Endothelial Function; Platelet Aggregation
Keywords: Secondhand smoke; passive smoking; platelet function; endothelial function

INTERVENTIONS:
Other: secondhand smoke exposure — Participants will be exposed to secondhand smoke for one hour. As a measure of secondhand smoke exposition, room carbon monoxide concentration will be continuously measured using an Ambient Carbon Monoxide Monitor APMA-360 and kept constant between 4.5-6.0 ppm. Levels in this magnitude are typically seen in smoking areas of restaurants and bars.

SUMMARY:
Passive smoking is associated with an increased risk for cardiovascular events. However, the exact mechanisms by which passive smoking affects cardiovascular health are not entirely understood. In the present study, the researchers investigate the effects of short-term exposure to secondhand smoke on platelet function and peripheral microvascular endothelial function in healthy individuals. For this purpose, platelet function and endothelial function are measured before and after a 1-hour exposure to secondhand smoke in a concentration that is encountered in bars and restaurants without smoke-free policies. The researchers' hypothesis is that short-term exposure leads to platelet activation and impairment of endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* nonsmokers
* no regular medication (in particular no drugs affecting platelet function or vascular function)

Exclusion Criteria:

* exposition to secondhand smoke within 1 week before inclusion
* use of drugs affecting platelet function or vascular function within 1 week before study inclusion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in platelet aggregation and/or endothelial function | 12-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Piero O. Bonetti, MD, Principal Investigator — Division of Cardiology, Department of Internal Medicine, Kantonsspital Graubuenden, Loestrasse 170, CH-7000 Chur, Switzerland
Locations (1):
- Kantonsspital Graubuenden, Chur, Switzerland